CLINICAL TRIAL: NCT01935180
Title: Does Cap Assisted Colonoscopy Improve Detection of Adenomatous Polyps? (CAP Trial)
Acronym: CAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Heiko Pohl, PI, White River Junction Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: DMS-22424
Record Dates: First submitted 2012-01-19; First posted 2013-09-04 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-08

CONDITIONS: Adenomatous Polyps
Keywords: colon polyps; adenoma resection; colon cancer screening; colonoscopy; polyp detection
MeSH Terms: conditions — Adenomatous Polyps; Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard colonoscopy (No Intervention)
- Cap assisted colonoscopy (Active Comparator): A transparent cap will be affixed to tip of the high-definition wide angle colonoscope.
  Interventions: Device: Colonoscopy Cap

INTERVENTIONS:
Device: Colonoscopy Cap — 4mm transparent cap (Olympus) mounted to the tip of a colonoscope.
  Arms: Cap assisted colonoscopy

SUMMARY:
Effectiveness of screening colonoscopy in cancer prevention relies on the detection and removal of adenomatous polyps. However, a substantial rate of adenomas is missed during a colonoscopy. It has been estimated that two thirds of missed adenomas are located on the proximal aspect of colonic folds. Attaching a transparent cap to the tip of a colonoscope may allow examination of the proximal aspect of colonic folds, and some early studies have suggested an increased polyp and adenoma detection using this technology. However, the studies have in part substantial methodological limitations (e.g. missing polyp histology, single endoscopist study, polyps not removed at the time of detection). Therefore, at this point it is unclear whether cap assisted colonoscopy may improve adenoma detection. The objective of this study is to evaluate whether cap assisted colonoscopy improves adenoma detection.

The investigators propose a two-center multiple endoscopists randomized controlled trial. Patients will be randomized to cap assisted colonoscopy or standard high definition white light colonoscopy. The cap is a 4mm commercially available transparent cap that is attached to the tip of the colonoscopy. Primary outcome measure is the adenoma detection rate (mean number of adenoma per patient). The investigators will assess and adjust for possible variables that can affect adenoma detection, including withdrawal time and quality of colon preparation. As a secondary outcome of interest the investigators will evaluate a possible learning curve effect among all endoscopists (a minimum of six) new to this method. In addition the investigators will evaluate whether cap assisted endoscopy improves real time prediction of polyp histology.

DETAILED DESCRIPTION:
All patients who present for a colonoscopy and meet inclusion and exclusion criteria will be asked to participate (see inclusion and exclusion criteria). All patients will undergo a regular bowel preparation with polyethylene glycol lavage (based on current standard of care) until clear rectal fluid is evacuated. Patients will be randomized to one of two groups:

1. Standard colonoscopy, or
2. Cap assisted colonoscopy. All colonoscopies will be performed using state of the art high-definition wide angle colonoscopy. The transparent cap, which is attached to the tip of the colonoscope, has a 4mm margin extending beyond the tip of the colonoscope. All patients will undergo a careful endoscopic examination. A timer will provide feedback on the time of insertion and the withdrawal time. Detected polyps will be assessed with standard white light and narrow band imaging to predict polyp histology (adenoma versus no adenoma), then resected and sent for histological evaluation according to standard of care. At least 8 experienced endoscopists at the participating centers will participate. Each endoscopist will perform at least 50 cap assisted colonoscopies as part of the study. Each endoscopist will be asked to complete a survey after 10 and after 50 cap assisted colonoscopies.

Patients will be randomized in blocks of four allocated to each examiner. The order of randomization will be computer generated. Information on randomization will be contained in sealed envelopes assigned to each examiner and individually opened immediately before the procedure after a patient's All participating endoscopist will fill out a questionnaire regarding the use of cap assistance colonoscopy after the initial 10 cap assisted colonoscopies and after at least 50 cap assisted cap colonoscopies. Endoscopists will also undergo a training session with respect to real time polyp diagnosis before study commencement and after each 20 colonoscopies enrollment.

ELIGIBILITY:
Inclusion Criteria:

• Any patient ≥ 50 years old and < 85 years old who presents for a colonoscopy with a potential for polyp resection and who does not meet any of the exclusion criteria mentioned below will be asked to participate

Exclusion criteria:

* Patients with known inflammatory bowel disease or active colitis
* Patients with familial adenomatous polyposis or other genetic syndromes that are associated with a high number of colonic polyps
* Patients who are receiving an emergency colonoscopy
* Poor general health (ASA class > 3)
* Patients on coumadin at the time of the procedure or with a coagulopathy and an elevated INR ≥ 1.5, or platelets < 50
* Patients who do not consent

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1148 (Actual)
Dates: Start 2010-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Pohl, Principal Investigator — White River Junction VAMC, Dartmouth Medical School
Locations (2):
- United States (2):
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - White River Junction VAMC, White River Junction, Vermont

REFERENCES:
- [Derived] von Renteln D, Kaltenbach T, Rastogi A, Anderson JC, Rosch T, Soetikno R, Pohl H. Simplifying Resect and Discard Strategies for Real-Time Assessment of Diminutive Colorectal Polyps. Clin Gastroenterol Hepatol. 2018 May;16(5):706-714. doi: 10.1016/j.cgh.2017.11.036. Epub 2017 Nov 23. PMID 29174789
- [Derived] von Renteln D, Robertson DJ, Bensen S, Pohl H. Prolonged cecal insertion time is associated with decreased adenoma detection. Gastrointest Endosc. 2017 Mar;85(3):574-580. doi: 10.1016/j.gie.2016.08.021. Epub 2016 Aug 31. PMID 27590962
- [Derived] Pohl H, Bensen SP, Toor A, Gordon SR, Levy LC, Berk B, Anderson PB, Anderson JC, Rothstein RI, MacKenzie TA, Robertson DJ. Cap-assisted colonoscopy and detection of Adenomatous Polyps (CAP) study: a randomized trial. Endoscopy. 2015 Oct;47(10):891-7. doi: 10.1055/s-0034-1392261. Epub 2015 Jun 30. PMID 26126162

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Colonoscopy: Standard colonoscopy without an attachment cap
Period: Overall Study
Arm/Group | Standard Colonoscopy | Cap Assisted Colonoscopy
Started | 573 | 575
Completed | 552 | 561
Not Completed | 21 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Colonoscopy | Cap Assisted Colonoscopy | Total
Number analyzed (Participants) | 552 | 561 | 1113
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (8.4) | 62.5 (8.3) | 61.8 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 209 | 195 | 404
  Male | 343 | 366 | 709
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 552 | 561 | 1113
Indication [Count of Participants; unit: Participants]
  Colonoscopy performed for cancer screening | 291 | 292 | 583
  Colonoscopy performed for polyp surveillance | 168 | 171 | 339
  Colonoscopy performed for symptoms (diagnostic) | 93 | 98 | 191

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Adenomas
Description: Mean number of adenomas per patient in each group.
Time Frame: duration of colonoscopy
Measure: Mean (Standard Deviation); unit: adenoma per patient
Groups:
- Standard Colonoscopy: Colonoscopy without a cap.
Arm/Group | Standard Colonoscopy | Cap Assisted Colonoscopy
Number analyzed (Participants) | 552 | 561
adenoma per patient | 0.82 (1.5) | 0.89 (1.6)

2. Secondary Outcome: Adenoma Detection Rate
Description: • Adenoma detection rate (ADR), % of patients with at least 1 adenoma
Time Frame: duration of colonoscopy
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Colonoscopy | Cap Assisted Colonoscopy
Number analyzed (Participants) | 552 | 561
Participants | 219 | 235

3. Secondary Outcome: Advanced Adenoma Detection Rate
Description: Proportion of patients with advanced adenomas
Time Frame: duration of colonoscopy
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Colonoscopy | Cap Assisted Colonoscopy
Number analyzed (Participants) | 552 | 561
Participants | 49 | 55

4. Secondary Outcome: Quality of Bowel Preparation
Description: Proportion of patients with a bowel preparation that was rated as good or excellent (four point scale that distinguishes the bowel prep as poor, fair, good or excellent).
Time Frame: duration of colonoscopy
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Colonoscopy | Cap Assisted Colonoscopy
Number analyzed (Participants) | 552 | 561
Participants | 518 | 502

5. Secondary Outcome: Withdrawal Time
Description: • Time taken for the withdrawal of the colonoscope from the cecum to anus among patients, who did not have any polyps.
Time Frame: time of colonoscope withdrawal
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Standard Colonoscopy | Cap Assisted Colonoscopy
Number analyzed (Participants) | 552 | 561
minutes | 8.9 [7.4 to 11.2] | 8.4 [6.7 to 10.2]

6. Secondary Outcome: Ease of Terminal Ileum Intubation
Description: • Proportion of patients, for whom intubation of the terminal ileum with the colonoscope was rated as "easy". Intubation could be rated by the endoscopist as "easy", "slightly difficult", "difficult", or "unable to intubate".
Time Frame: during colonoscopy
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Colonoscopy | Cap Assisted Colonoscopy
Number analyzed (Participants) | 552 | 561
Participants | 435 | 473

7. Secondary Outcome: Real Time Prediction of Polyp Histology
Description: Difference in recommended surveillance interval between real time polyp diagnosis and pathological diagnosis among patients with at least one diminutive polyp
Time Frame: duration of colonoscopy
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Colonoscopy | Cap Assisted Colonoscopy
Number analyzed (Participants) | 269 | 297
Participants | 246 | 281

ADVERSE EVENTS:
Arm/Group | Standard Colonoscopy | Cap Assisted Colonoscopy
Serious Adverse Events (participants affected / at risk) | 0/552 | 0/561
Other Adverse Events (participants affected / at risk) | 0/552 | 0/561

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No